CLINICAL TRIAL: NCT06533306
Title: Estimation of the Risk of Presenting Metachronous Acquired Contralateral Cryptorchidism in Patients With a History of Unilateral Cryptorchidism.
Brief Title: Metachronous Acquired Contralateral Cryptorchidism in Patients With a History of Unilateral Cryptorchidism.
Status: Completed | Type: Observational
Sponsor: Consorci Sanitari de l'Alt Penedès i Garraf (Other)
Responsible Party: Sponsor
Other Study IDs: CSAPG-63
Record Dates: First submitted 2024-07-25; First posted 2024-08-01 (Actual); Last update posted 2024-08-01 (Actual); Status verified 2024-07

CONDITIONS: Cryptorchidism
Keywords: Cryptorchidism
MeSH Terms: conditions — Cryptorchidism | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Surgery for cryptorchidism. — Patients previously operated on for cryptorchidism.

SUMMARY:
The present study aims to calculate the risk of a patient with a history of cryptorchidism developing cryptorchidism on the contralateral side.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 13 years or older, previously operated on for cryptorchidism.

Exclusion Criteria:

* Diagnosis of endocrine disease or any polymalformative syndrome.
* Synchronous bilateral cryptorchidism.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients previously operated on for cryptorchidism
Sampling Method: Non-Probability Sample
Enrollment: 126 (Actual)
Dates: Start 2024-04-01 (Actual); Primary Completion 2024-05-30 (Actual); Study Completion 2024-05-30 (Actual)

PRIMARY OUTCOMES:
Contralateral Cryptorchidism | Up to 1 month
  Proportion of patients previously operated on for cryptorchidism in whom acquired contralateral cryptorchidism is detected.

CONTACTS AND LOCATIONS:
Overall Officials: Carme Grande Moreillo, MD, Principal Investigator — CSAPG
Locations (1):
- Consorci Sanitari Alt Penedès-Garraf, Vilafranca del Penedès, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Yes
IPD (without personal identification data) could be shared by requirement from other researchers after the end of the study, and only for research purposes and previous approval of promotor center of the study (CSAPG). Anyway, Spanish and European Union legal policy about data protection will strictly be followed (IPD will not be transferred outside European Union).
Supporting Information: Study Protocol
Time Frame: After publication of main results of the study.
Access Criteria: IPD will be shared only for scientific research purposes and following the Spanish and European Union normative law about data protection. The requirements will be directed to the IP of the study. The IP will evaluate the request to verify and evaluate the data that is requested and the purposes for which it is requested. Next, the IP will transfer the request to the promotor center the study for the final decision.